CLINICAL TRIAL: NCT07300722
Title: Impact of "SI Kumbang" Gymnastic Exercise on Physical Performance and Immunity in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umi Sjarqiah (Other)
Collaborators: Fakultas Kedokteran dan Kesehatan Universitas Muhammadiyah Jakarta (Other); Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor-Investigator, Umi Sjarqiah, Medical Doctor, Universitas Muhammadiyah Yogyakarta
Organization: Universitas Muhammadiyah Yogyakarta (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24-10-1593
Record Dates: First submitted 2025-11-19; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: physical performance; immunity; SI Kumbang exercise gymnastics; elderly

STUDY DESIGN:
Intervention Model Description: The SI Kumbang gymnastics exercise and Bugar Lansia gymnastics exercise regimens were part of the intervention groups. For 12 weeks in a row, both therapies included three 30-minute sessions, 3 times per week. Participants received adaption sessions to acquaint themselves with the workout regimens throughout the first week. The Borg Scale was utilized to track intensity.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SI Kumbang Gymnastic Exercise (Experimental): Intervention Group received SI Kumbang gymnastic exercise
  Interventions: Other: SI Kumbang gymnastic exercise
- Bugar Lansia Gymnastic Exercise (Active Comparator): Controlled Group received Bugar Lansia gymnastic exercise
  Interventions: Other: Bugar Lansia Gymnastic Exercise

INTERVENTIONS:
Other: SI Kumbang gymnastic exercise — SI Kumbang Gymnastic Exercise with four-way leg movements with hand movements using barbell weights and medium-intensity music.
  Arms: SI Kumbang Gymnastic Exercise
Other: Bugar Lansia Gymnastic Exercise — Bugar Lansia Gymnastic Exercise with one-way forward leg movements with hand movements without barbell weights with medium intensity music.
  Arms: Bugar Lansia Gymnastic Exercise

SUMMARY:
The goal of this clinical trial is to evaluate and compare the impact of SI Kumbang gymnastic exercise and Bugar Lansia gymnastic exercise programs on physical performance dan immunity in elderly. It will also learn about the safety of SI Kumbang gymnastic exercise. The main questions it aims to answer are:

* How does cardiorespiratory fitness differ between SI Kumbang and Bugar Lansia exercise?
* How does muscle strength differ between SI Kumbang and Bugar Lansia exercise?
* How does balance differ between SI Kumbang and Bugar Lansia exercise?
* How does physical activity differ between SI Kumbang and Bugar Lansia exercise?
* How do Caspase-1 and IL-18 inflammasomes differ between SI Kumbang and Bugar Lansia exercise? Researchers will compare SI Kumbang gymnastic exercise to a Bugar Lansia gymnastic exercise to see if SI Kumbang gymnastic exercise better than Bugar Lansia gymnastic exercise.

Participants will:

* Do SI Kumbang gymnastic exercise or Bugar Lansia gymnastic exercise a within 3 times a week for 3 months.
* Visit the clinic twice for outcome assesment before and after intervention.
* Keep a diary of their symptoms.

DETAILED DESCRIPTION:
A sample size of 33 people per group was determined. The study supervisor oversaw the use of a basic randomization program to carry out the random allocation. The Sequentially Numbered, Opaque, Sealed Envelope (SNOSE) technique was used to guarantee allocation concealment. Outcome assessors were subjected to single blinding; they were not told about group allocations and were not allowed to look for relevant information. The "SI Kumbang" and "Bugar Lansia" gymnastics exercise regimens were part of the intervention groups. For 12 weeks in a row, both therapies included three 30-minute sessions per week. Participants received adaption sessions to acquaint themselves with the workout regimens throughout the first week. The Borg Scale was utilized to track intensity.

The research team reviewed patient logbooks at the beginning of each week to track adverse effects such weariness, shortness of breath, pain, or dizziness. At RS Islam Jakarta Pondok Kopi, every suspected adverse event was swiftly assessed, and any required medical attention was given. Every adverse event was reported to the ethics committee of the institution.

Data analysis was performed using SPSS 29.0 tests with significance set at p<0.05. Descriptive summaries of the sample characteristics were provided. Prior to analysis, the normality of the data was checked. Dependent t-tests were used to compare pre intervention and post intervention score in the SI Kumbang and Bugar Lansia groups for normally distributed outcomes (6MWD, handgrip, SPPB, PASE, Caspase-1, IL-18); the Wilcoxon test was used to assess non-normal data. Independent t test or Mann-Whitney U test is used for compared the effectiveness of the two interventions (∆ score). A p-value of less than 0.05 was deemed significant.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Age of 60 to 70 years old.
* Categorized as pre-frail (FI-40 score > 0.08 < 0.25) or robust (FI-40 score ≤ 0.08)
* Body mass index (BMI) between 18.5 and 24.9.
* Diabetes mellitus (controlled glucose ≤ 120 mg/dL)
* Blood pressure (controlled blood tension ≤ 130/80 mmHg) without taking any drugs that affected heart rate.

Exclusion Criteria:

* Chronic heart or lung disease conditions
* Chronic conditions that cannot be reversed (e.g., cancer or chronic renal disease)
* Diabetes complications in the extremities
* Motor impairment (MMT < 5)
* Knee pain
* Lower limb deformities (genu varus/valgus)
* Hand deformities

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiration endurance as Assessed by Six-Minute Walk Distance (6MWD) | From enrollment to the end of treatment at 12 weeks.
  The definition of Six Minute Walking Distance (6MWD) is a 15-meter walking test for 6 minutes which is one of the sub-maximal tests, namely O2 uptake and heart rate are linearly related to VO2max so that fitness can be predicted. During the exercise, respondents are not allowed to run and respondents are allowed to rest during the test. This is an appropriate method because it has been proven to be able to achieve the sub-maximal zone and aerobic zone in a person. The results taken are the distance traveled in meters (Six Minutes Walking Distance).
Strength muscle as Assessed by handgrip JAMAR | From enrollment to the end of treatment at 12 weeks.
  A Jamar is a handheld dynamometer used to measure the maximal strength of the hand and forearm muscles through an isometric grip test. It assesses the strength of the muscles primarily responsible for closing the fingers and gripping, such as the forearm flexors. The test involves a standardized procedure, and the results are displayed on a dual scale in kilograms and pounds, often with a peak-hold needle to record the highest force achieved.
Balance as Assessed by Short Physical Performance Battery (SPPB). | From enrollment to the end of treatment at 12 weeks
  The Short Physical Performance Battery (SPPB) is an objective assessment tool used to evaluate the physical function of an older person's lower extremities. It is comprised of three simple tasks: a timed chair stand test, a timed gait speed test, and a standing balance test. The results from these tests are combined into a score from 0 (worst) to 12 (best), which is used to predict various health outcomes such as disability, hospitalization, and mortality.
Physical activity as Assessed by Physical Activity Scale for the Elderly (PASE). | From enrollment to the end of treatment at 12 weeks.
  The Physical Activity Scale for the Elderly (PASE) is a brief, self-report questionnaire that assesses the level of physical activity in adults aged 65 and older over a one-week period. It includes questions about frequency and duration of leisure, household, and work-related activities and can be administered through telephone, mail, or in-person interviews. Higher scores indicate a greater amount of physical activity.
Immunity were inflammasome as Assessed by Caspase-1 and IL-18. | From enrollment to the end of treatment at 12 weeks.
  Caspase-1 is an enzyme that activates the proinflammatory cytokines interleukin-1 beta (IL-1β) and interleukin-18 (IL-18) by processing them into their mature, active forms. This process is a key part of the body's inflammatory response to infections and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Umi Sjarqiah, Medical Doctor, Principal Investigator — University of Muhammadiyah Jakarta
Locations (1):
- University of Muhammadiyah Jakarta, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT07300722/Prot_SAP_000.pdf